CLINICAL TRIAL: NCT06954623
Title: Partial Breast Re-irradiation for Breast Cancer Recurrences After Repeat Breast-conserving Surgery With Proton Beam Therapy
Brief Title: Partial Breast Re-irradiation for Breast Cancer
Acronym: BREAST
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital Heidelberg (Other)
Responsible Party: Principal Investigator, Juergen Debus, Head of Department Radiation Oncology, University Hospital Heidelberg
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RADONK-2024-BREAST
Record Dates: First submitted 2025-04-16; First posted 2025-05-01 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Breast Cancers
Keywords: re-irratdiation; proton beam
MeSH Terms: conditions — Breast Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Proton beam therapy (Experimental)
  Interventions: Radiation: Radiation Therapy

INTERVENTIONS:
Radiation: Radiation Therapy — proton beam radiation

SUMMARY:
Breast cancer is the most common malignancy in women. Breast-conserving surgery (BCS) with adjuvant whole-breast irradiation (WBI) is currently the standard of care in the oncological treatment of primary breast cancer and offers an equivalent alternative to mastectomy. The primary aim of adjuvant radiotherapy (RT) is to improve local control and thus improve overall survival and breast cancer-specific mortality. However, nodal-negative women have a 10-year risk for local recurrences after RT in up to 15.6%. The management of ipsilateral breast cancer recurrence depends on the extent of tumor disease and staging results at the time of recurrence and mastectomy is currently the standard of care for previously irradiated patients. The application of particle therapy using proton beam therapy (PBT) represents an innovative radiotherapeutic technique for breast cancer patients. This trial will be conducted as a prospective single-arm phase II study in 20 patients with histologically proven invasive breast cancer recurrences with negative margins after repeat BCS and with an indication for local re-irradiation. Required time interval will be 1 year after previous RT to the ipsilateral breast. Patients will receive partial breast re-RT with proton beam therapy in 15 once daily fractions up to a total dose of 40.05 GyRBE. The primary endpoint is defined as the cumulative overall occurrence of acute / subacute skin toxicity grade ≥3 within 6 months after the start of re-RT.

DETAILED DESCRIPTION:
The therapeutic challenge in re-irradiation involves finding a balance between tumor control and the risk of severe toxicity from cumulative radiation doses in previously irradiated organs. Re-RT options include the use of brachytherapy (BT) ], intraoperative radiotherapy (IORT) or external beam RT with photons or electrons. Depending on the time interval since previous RT and applied technique, high-grade (≥3) toxicity rates for re-RT range from about 9% acute skin to 12 % - 17 % late fibrosis and 1% - 10 % G4 toxicity for BT, late grade 3 fibrosis of 21% for IORT and grade 3 toxicity (skin, esophagitis, wound dehiscence) of 7 - 24% - 35% for EBRT including late breast volume asymmetry in 12%, acute and late grade 4 ulceration (1-2%) and even grade 5 (treatment related deaths) in 1.2%.

The dosimetric profile of PBT with the Bragg Peak offers advantageous physical properties and has proven to be superior to photon-based techniques in respect of dose reduction to adjacent organs-at-risk (OAR) and effective target volume coverage with lower integral doses to the patient's whole body. In addition, this technique could potentially offer higher radiobiological effects and tumor responses [28], which is particularly advantageous in potentially more therapeutically resistant disease biology in breast cancer recurrences. Overall, prospective experience related to re-RT of the ipsilateral breast after recurrences is limited and most commonly involves the technique of invasive multicatheter brachytherapy.

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed recurrent (or new primary) ipsilateral invasive breast cancer or DCIS after prior RT of the ipsilateral breast
* indication for re-irradiation after repeat breast conserving surgery (e.g. lumpectomy, wide excision, …)
* tumor size < 3 cm
* clinically node-negative (cN0)
* negative resection margin (R0)
* time interval: start of re-RT to prior RT ≥ 12 months
* ECOG Performance status ≤ 2
* ability of subject to understand character and individual consequences of the clinical trial
* written informed consent
* ≥18 years of age

Exclusion Criteria:

* distant metastases

  * concomitant chemotherapy (concomitant endocrine hormonal therapy is allowed; sequential chemotherapy is allowed)
  * patients who have not recovered from acute toxicities of prior therapies
  * known carcinoma < 5 years ago (excluding Carcinoma in situ of the cervix, basal cell carcinoma, squamous cell carcinoma of the skin) requiring immediate treatment interfering with study therapy
  * pregnant or lactating women
  * participation in another competing clinical study or observation period of competing trials
  * history of active connective tissue disorder (i.e. systemic lupus erythematosus, scleroderma, dermatomyositis, xeroderma pigmentosum, …)
  * medical implants, which are at the time of reirradiation not eligible for particle therapy at Heidelberg Ion Beam Therapy Center

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 20 (Estimated)
Dates: Start 2025-08-28 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2029-09-01 (Estimated)

PRIMARY OUTCOMES:
skin toxicity | Within the first 6 months after the start of re-RT
  Occurrence of overall acute / subacute skin toxicity CTCAE grade 3 or higher (NCI CTCAE version 5.0) assessed.

SECONDARY OUTCOMES:
Local Tumor control | At 1, 2 and 5 years after re-RT
  presence of tumor cells on initial tumor site
Patients Quality of life | At 1, 2 and 5 years after re-RT
  quality of life (EORTC QLQ-C30 and the supplementary questionnaire module QLQ-BR42 measuring specific quality of life aspects related to breast cancer treatment)
Regional Tumor control | At 1, 2 and 5 years after re-RT
  presence of tumor cells on initial tumor region
Distant Tumor control | At 1, 2 and 5 years after re-RT
  presence of tumor cells on distant tumor site
progression-free survival | At 1, 2 and 5 years after re-RT
  patients without a tumorprogress
overall survival | At 1, 2 and 5 years after re-RT
  alive patients
Quality of life -C30 | At 1, 2 and 5 years after re-RT
  scores ranging from 0 to 100, with 0 being the lowest score
Quality of life BR-42 | At 1, 2 and 5 years after re-RT
  Scores ranging from 0 to 100, 0 being the lowest score

CONTACTS AND LOCATIONS:
Overall Officials: Juergen Debus, MD, Principal Investigator — University Hospital Heidelberg
Locations (1):
- University Hospital Heidelberg, Department Radiation Oncology, Heidelberg, Germany

IPD SHARING:
Plan to Share IPD: No